CLINICAL TRIAL: NCT02301650
Title: The Effect of Anti-viral Drugs Used in Late Pregnancy in Mothers With Hepatitis B Virus Infection on Long-term Development of Children
Brief Title: The Effect of Anti-viral Drugs Used in Late Pregnancy on Long-term Development of Children
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Wei Yi, Chief physician, Beijing Ditan Hospital
Other Study IDs: Z141107002514131
Record Dates: First submitted 2014-11-12; First posted 2014-11-26 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: the Safety of Anti-viral Drugs Used in Late Pregnancy
Keywords: Hepatitis B virus; pregnancy; nucleoside (acid) analogs; children; safety
MeSH Terms: conditions — Hepatitis B; Heartburn | interventions — Lamivudine; Telbivudine; Tenofovir

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- group A: The one year old children born in Beijing Ditan hospital and whose mothers had taken Lamivudine in late pregnancy
  Interventions: Drug: Lamivudine
- group B: The one year old children born in Beijing Ditan hospital and whose mothers had taken Telbivudine in late pregnancy
  Interventions: Drug: Telbivudine
- group C: The one year old children born in Beijing Ditan hospital and whose mothers had taken Tenofovir in late pregnancy
  Interventions: Drug: Tenofovir
- group D: The one year old children born in Beijing Ditan hospital and whose mothers untreated in late pregnancy

INTERVENTIONS:
Drug: Lamivudine — mothers use Lamivudine in late pregnancy
  Other Names: 3-TC; CAS: 134678-17-4
  Groups: group A
Drug: Telbivudine — mothers use Telbivudine in late pregnancy
  Other Names: CAS: 3424-98-4
  Groups: group B
Drug: Tenofovir — mothers use Tenofovir in late pregnancy
  Other Names: Tenofovir Disoprox; CAS: 147127-20-6
  Groups: group C

SUMMARY:
Mother to child transmission(MTCT) is the main route of hepatitis B virus(HBV) transmission.High HBV DNA level of pregnant women is the main risk factor of MTCT. Many literatures demonstrate that using nucleoside (acid) analogs in late pregnancy can significantly reduce HBV DNA level and effectively blocking MTCT. Therefore, treatment guidelines of hepatitis B in Europe and the Asia Pacific region clearly pointed out: Nucleoside (acid) analogs can be used in pregnant women after 28 weeks of gestation for blocking MTCT in mothers with high HBV DNA level. At present, the drugs used in late pregnancy including lamivudine (LAM) ,telbivudine(LdT) and tenofovir(TDF).

The safety of nucleoside (acid) analogues used in late pregnancy on children is not clear.In most of the related researches,the observation termination was 7-12 months after birth, and most were concentrated on the blocking effect of MTCT.The long-term impact of Nucleoside (acid) analogues on children's development has not been reported in the literatures. The aim of this study is to make clear of the effect of nucleoside (acid) analogues used in late pregnancy on long-term impact of children's development.

The one year old children born in Beijing Ditan hospital and whose mothers had taken LAM,LdT or TDF during late pregnancy will be enrolled as study group, and eligible children whose mothers untreated will be enrolled as control group. The children's height, weight, nutritional status, developmental quotient and immune response to hepatitis B vaccine etc will be evaluated at baseline and at 3 years old. By comparing the children's development in different groups as well as in self-control of different ages, we will discuss the effect of Nucleoside (acid) analogues on children's long-term development.

ELIGIBILITY:
Inclusion Criteria:

* The one year old children whose mothers had taken Lamivudine,Telbivudine or Tenofovir in late pregnancy(28-30 weeks of gestation);
* The one year old children whose mothers untreated in late pregnancy;
* Children had completed standard hepatitis B vaccine and hepatitis B immune globulin combined active and passive prophylaxis;
* HBV DNA level of the children's mothers were over 6.0 log10 IU/ml before 28 weeks of gestation.

Exclusion Criteria:

* Children whose mothers over 35 years old at delivery;
* The couple having family hereditary disease or abnormal malformation has been found at fetal screening before 28 weeks gestation;
* History of amniocentesis during pregnancy;
* Co-infection with either hepatitis C virus, hepatitis D virus, human immunodeficiency virus, syphilis, toxoplasmosis, rubella or cytomegalovirus.
* Complications of pregnancy-induced hypertension, premature rupture of membranes, preterm birth, placenta previa or placental abruption; asphyxia at birth.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The one year old children born in BeiJing DiTan Hospital and whose mothers had taken Lamivudine, Telbivudine or Tenofovir and untreated in late pregnancy with HBV DNA level over 6.0 log10 IU/ml
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The rate of abnormal development | 6 months
  The children' development will be measured by Gesell Developmental Scales, including adaptability, mobility, fine motion skills, language ability and social skills.The children will be considered normal if the score is ≥86, score between 76-85 is suspicious, and score≤75 is abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Yi, Principal Investigator — Beijing Ditan Hospital